CLINICAL TRIAL: NCT00552513
Title: An International Randomised Trial of Early Versus Delayed Invasive Strategies in Patients With Non-ST Segment Elevation Acute Coronary Syndromes
Brief Title: Early Versus Delayed Timing of Intervention in Patients With Acute Coronary Syndromes
Acronym: TIMACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FRN: MCT-79654; ISRCTN20993046 (Registry Identifier: International Standard Randomised Controlled Trial Number)
Record Dates: First submitted 2007-10-30; First posted 2007-11-02 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Unstable Angina; Myocardial Infarction
Keywords: timing; intervention; early; delayed; acute coronary syndromes; PCI; angiography; Non ST-segment elevation myocardial infarction; unstable angina
MeSH Terms: conditions — Angina, Unstable; Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Coronary Intervention (Other): Coronary angiography and intervention (either percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG] surgery) as soon as possible (within 24 hours of randomisation).
  Interventions: Procedure: Early Coronary Intervention
- Delayed Coronary Intervention (Other): Delayed intervention: Coronary angiography and intervention (either percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG] surgery) any time after 36 hours after randomisation.
  Interventions: Procedure: Delayed Coronary Intervention

INTERVENTIONS:
Procedure: Early Coronary Intervention — Perform coronary angiography and intervention (either percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG] surgery) as soon as possible (and within 24 hours of randomisation).
  Arms: Early Coronary Intervention
Procedure: Delayed Coronary Intervention — Perform coronary angiography and intervention (either percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG] surgery) any time after 36 hours after randomisation.
  Arms: Delayed Coronary Intervention

SUMMARY:
The timing of intervention study is a prospective, randomized, international, multicentre comparison of the relative efficacy, safety, and cost effectiveness of a management strategy of coronary angiography and intervention performed within 24 hours of randomization versus delayed coronary angiography and intervention in patients after 36 hours with acute coronary syndromes (ACS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting or admitted to hospital with symptoms suspected to represent an acute coronary syndrome (unstable angina or MI without persistent ST elevation) i.e., clinical history consistent with new onset, or a worsening pattern, of characteristic ischemic chest pain or ischemic symptoms occurring at rest or with minimal activity (lasting longer than five minutes or requiring sublingual nitroglycerin for relief of the pain)
2. Able to randomise within 24 hours of the onset of the most recent episode of symptoms
3. At least two of the three following additional criteria:

   * Age more than or equal to 60 years
   * Troponin T or I or Creatine Kinase - Myocardial Bands (CK-MB) above the upper limit of normal for the local institution
   * ElectroCardioGram (ECG) changes compatible with ischemia (i.e., ST depression at least 1 mm in two contiguous leads or T wave inversion mroe than 3 mm or any dynamic ST shift or transient ST elevation)
4. Written informed consent dated and signed

Exclusion Criteria:

1. Age less than 21 years
2. Not a suitable candidate for revascularisation
3. Co-morbid condition with life expectancy less than six months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3031 (Actual)
Dates: Start 2005-05; Primary Completion 2008-07 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shamir Mehta, MD, MSc, Principal Investigator — Population Health Research Institute, Hamilton Health Sciences, McMaster University
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Background] MICHELANGELO OASIS 5 Steering Committee; Mehta SR, Yusuf S, Granger CB, Wallentin L, Peters RJ, Bassand JP, Budaj A, Joyner C, Chrolavicius S, Fox KA. Design and rationale of the MICHELANGELO Organization to Assess Strategies in Acute Ischemic Syndromes (OASIS)-5 trial program evaluating fondaparinux, a synthetic factor Xa inhibitor, in patients with non-ST-segment elevation acute coronary syndromes. Am Heart J. 2005 Dec;150(6):1107. doi: 10.1016/j.ahj.2005.09.025. PMID 16338245
- [Result] Mehta SR, Granger CB, Boden WE, Steg PG, Bassand JP, Faxon DP, Afzal R, Chrolavicius S, Jolly SS, Widimsky P, Avezum A, Rupprecht HJ, Zhu J, Col J, Natarajan MK, Horsman C, Fox KA, Yusuf S; TIMACS Investigators. Early versus delayed invasive intervention in acute coronary syndromes. N Engl J Med. 2009 May 21;360(21):2165-75. doi: 10.1056/NEJMoa0807986. PMID 19458363
- See also: Population Health Research Institute — http://www.phri.ca

RESULTS

PARTICIPANT FLOW:
Groups:
- Early: Coronary angiography and intervention (either percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG] surgery) as soon as possible (within 24 hours of randomisation).
- Delayed: Delayed intervention: Coronary angiography and intervention (either percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG] surgery) any time after 36 hours after randomisation.
Period: Overall Study
Arm/Group | Early | Delayed
Started | 1593 | 1438
Completed | 1588 | 1437
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early | Delayed | Total
Number analyzed (Participants) | 1593 | 1438 | 3031
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 65.1 (0) | 65.8 (0) | 65.5 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 554 | 498 | 1052
  Male | 1039 | 940 | 1979

OUTCOME MEASURES:

1. Primary Outcome: Composite of Death, Myocardial (re-) Infarction, or Stroke
Time Frame: 180 days
Population: All patients were included in the final intention-to-treat analysis. Event rates in the two groups were estimated with the use of the Kaplan-Meier method. The hazard ratio and two-sided 95% confidence intervals were calculated with the use of a Cox proportional-hazards model.
Measure: Number; unit: participants
Groups:
- Early Intervention: Coronary angiography to be performed as rapidly as possible and within 24 hours after randomization
- Delayed Intervention: Coronary angiography to be performed after a minimum delay of 36 hours after randomization
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 1593 | 1438
participants | 153 [0.68 to 1.06] | 163 [0.68 to 1.06]
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; Test type: Superiority or Other; p = 0.15, Regression, Logistic; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.68 to 1.06]

2. Secondary Outcome: First Occurrence of Any Component of the Composite of Death, MI, or Refractory Ischemia
Time Frame: 180 days
Measure: Number; unit: participants
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 1593 | 1438
participants | 151 | 186
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; Test type: Superiority or Other; p = 0.003, Regression, Logistic; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.58 to 0.89]

3. Secondary Outcome: Composite of Death, MI, Stroke, Refractory Ischemia or Repeat Revascularization at 180 Days
Time Frame: 180 days
Measure: Number; unit: Eparticipants
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 1593 | 1438
Eparticipants | 264 | 280
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; Test type: Superiority or Other; p = 0.04, Regression, Logistic; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.71 to 0.99]

4. Secondary Outcome: Stroke at 30 Days and 180 Days
Time Frame: 180 days
Reporting Status: Not Posted

5. Secondary Outcome: Need for Mechanical or Pharmacological Coronary Revascularization (i.e. Thrombolysis, PCI, CABG) at Days 30, 90, and 180
Time Frame: 180 days
Reporting Status: Not Posted

6. Secondary Outcome: In-hospital Major Bleeding
Time Frame: Hospital discharge
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Early | Delayed
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PHRI agreements may vary with individual investigators, but will not prohibit any investigator from publishing. PHRI supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.